CLINICAL TRIAL: NCT06567977
Title: TriMaximize: A Multicentre, Prospective, Non-interventional Trial Monitoring Therapy Pathways of Asthma Patients Treated With an Extra-fine ICS/LABA/LAMA Single-inhaler Triple Therapy in a Real-world Setting and Characterizing the Effects on Health-related Outcomes.
Brief Title: TriMaximize: A Multicentre, Prospective, Non-interventional Trial in Asthma Patients
Acronym: Trimaximize PL
Status: Recruiting | Type: Observational
Sponsor: Chiesi Poland Sp. z o.o. (Industry)
Collaborators: Gesellschaft für Therapieforschung mbH (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS 005 Pn
Record Dates: First submitted 2024-03-05; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Trimbow — Trimbow® is a fixed triple therapy containing a long-acting muscarinic antago-nist (LAMA, Glycopyrronium), a long-acting beta-adrenergic agonist (LABA, Formoterol) and an inhaled corticosteroid (ICS, beclomethasone). Trimbow® has an extra-fine formulation delivered as a controlled dosage aerosol. Trim-bow® is to be applied in accordance with its current marketing authorisation and the guidance specified in the summary of product characteristics (SmPC) in each country.
  Other Names: Trimbow®

SUMMARY:
TriMaximize: A multicentre, prospective, non-interventional trial monitoring therapy pathways of asthma patients treated with an extra-fine ICS/LABA/LAMA single-inhaler triple therapy in a real-world setting and characterizing the effects on health-related outcomes.

DETAILED DESCRIPTION:
The goals of asthma therapy for all degrees of disease severity are minimising asthma symptoms, maximising lung function, and preventing asthma exacer-bations. Despite the existing treatment options and differentiated guidelines, 35 % to 45 % of the GINA 4/5 patients suffer from inadequately controlled symptoms. To investigate the cause of unsatisfactory treatment results, it is essential to monitor therapy pathways of asthma patients in a real-world set-ting. Resulting data can be compared to therapy guidelines and generate hy-potheses for future clinical trials.

Trimbow® is a fixed triple therapy containing a long-acting muscarinic antago-nist (LAMA, glycopyrronium), a long-acting beta-adrenergic agonist (LABA, formoterol) and an inhaled corticosteroid (ICS, beclomethasone). Trimbow® MS (medium strength) contains 100 µg beclomethasone whereas Trimbow® HS (high strength) contains 200 µg beclomethasone. Both formulations are investigated in this study.

Trimbow® has shown major clinical benefits in randomised controlled trials. However, the effects of Trimbow® on changes in patients' symptom burden and quality of life, adherence and clinical outcomes have not been yet as-sessed in a real-world asthma patient population.

The primary objective is to describe patient characteristics and therapy path-ways for patients with a diagnosis of moderate to severe asthma who are treated with Trimbow® in real world practice.

Secondary objectives include:

* To assess asthma control (ACT)
* To assess quality of life (Mini-AQLQ)
* To assess treatment adherence (TAI)
* To analyse parameters of lung function
* To analyse parameters of small airways disease (FEF 25-75, RV/TLC)
* To analyse parameters of asthma-related airway inflammation (FeNO)
* To analyse parameters of persistent airways limitation (reversibility testing FEV1/FVC)
* To analyse the incidence and the severity of asthma exacerbations
* To analyse the use of rescue medication
* To analyse the use of systemic corticosteroids
* To assess healthcare resource utilisation
* To assess treatment satisfaction with Trimbow®
* To assess tolerability of Trimbow® This is a non-interventional, longitudinal, international, multicentre study with prospective data collection. At baseline, the patient's medical history with spe-cial focus on asthma will be collected. The study baseline visit is at the time point of start of treatment with Trimbow®. Trimbow® treatment may have started up to a maximum of 4 weeks prior to inclusion of the patient into this NIS.

The planned observational period per patient should be at least 52 weeks (ob-servational period [OP] I of the study) and can be extended to up to 3 years (OP II of the study). During the observational period, data may be collected approximately every 3 months during the first year (OP I of the study) and thereafter every 6 months (OP II of the study). The present observational plan does not stipulate any study-related procedures or defined time points; only data that are available within the current clinical routine will be collected as documented in the patients' files.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age,
* Patients with confirmed leading diagnosis of asthma with or without concomitant COPD,
* Physician decision to start fixed triple therapy with ICS/LABA/LAMA (Trimbow® MS or HS) according to its current authorised indication. The treatment decision must be made independently from participation in this NIS,
* Patients willing and able to sign an informed consent for use of their pseudonymised clinical data within the present non-interventional study.

Exclusion Criteria:

• Participation in an interventional clinical trial within 30 days prior to en-rolment into the present non-interventional study or planned enrolment in an interventional clinical trial during the observational period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult asthmatic patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to describe patient characteristics and therapy path-ways for patients with a diagnosis of moderate to severe asthma who are treated with Trimbow in real world practice. | 12 months
  Primary outcome measures include:
  Descriptive analisys of patients demografic
  Descriptive analisys of patient demographic

SECONDARY OUTCOMES:
Assess asthma control (ACT) | 12 months
  - Assess asthma control (ACT) - Change from baseline in ACT scores
Assess quality of life To measure the functional impairments | 12 months
  - Assess quality of life - Change from baseline in Mini-AQLQ scores
Treatment adherence | 12 months
  - Assess treatment adherence - Change from baseline in TAI scores
Lung function | 12 months
  - Analyse parameters of lung function using spirometry - Change from baseline in FEV1
Small airways parameters | 12 months
  - Analyse parameters of small airways disease - Change from baseline in small airway function measured by pre-dose AUCAX (Area under the curve of reactance) using available oscillometry system
Airway inflammation | 12 months
  - Analyse parameters of asthma-related airway inflammation - Change from baseline in percentage of patients with a fraction of exhaled nitric oxide (FeNO) below or above 20 ppb
Persistent airflow limitation | 12 months
  - Analyse parameters of persistent airflow limitation - Change from baseline in percentage of patients with persistent airflow limitation (PAL); PAL defined as post-BD FEV1 <80% predicted and post-BD FEV1/FVC Ratio < 0.7
Asthma exacerbations | 12 months
  - Analyse the incidence of asthma exacerbations - Number of exacerbations 12 months prior to baseline and during study
Rescue medication use | 12 months
  - Analyse use of rescue medication - Use of any rescue medication 7 days prior to baseline and during study 7 days prior to respective visit
Systemic corticosteroids use | 12 months
  - Analyse use of systemic corticosteroids - Use of any systemic corticosteroids 12 months prior to baseline and during study
Adverse events occurence | 12 months
  - Assess adverse events associated with use of Trimbow - Assessment of the number and type of adverse events
Retention rate with Trimbow | 12 months
  - Assess retention rate with Trimbow - Assess continuation of treatment with Trimbow (retention rate of Trimbow) at month 12

CONTACTS AND LOCATIONS:
Locations (1):
- Indywidualna Specjalistyczna Praktyka Lekarska, Tarnowskie Góry, Poland

IPD SHARING:
Plan to Share IPD: No